CLINICAL TRIAL: NCT02760797
Title: An Open-Label, Multicenter, Dose-Escalation Phase Ib Study With Expansion Phase to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Therapeutic Activity of Emactuzumab and RO7009789 Administered in Combination in Patients With Advanced Solid Tumors
Brief Title: A Study of Emactuzumab and RO7009789 Administered in Combination in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP29427; 2015-004348-21 (EudraCT Number)
Record Dates: First submitted 2016-04-14; First posted 2016-05-04 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — emactuzumab; selicrelumab

ARMS (2):
- Part I (Dose-Finding Stage) (Experimental): Emactuzumab and RO7009789 will be administered intravenously (IV) at a starting dose of 500 milligrams (mg) for emactuzumab and 2 mg for RO7009789. Treatment will continue as long as there is clinical benefit until unacceptable toxicity, symptomatic deterioration, or withdrawal of consent.
  Interventions: Drug: Emactuzumab; Drug: RO7009789
- Part II (Dose Expansion Stage) (Experimental): Emactuzumab and RO7009789 will be administered IV at the maximum tolerated dose defined in Part I of the study. Treatment will continue as long as there is clinical benefit until unacceptable toxicity, symptomatic deterioration, or withdrawal of consent.
  Interventions: Drug: Emactuzumab; Drug: RO7009789

INTERVENTIONS:
Drug: Emactuzumab — Emactuzumab will be administered IV every 3 weeks (every cycle) during Part I and every 3 or 6 weeks (every cycle or every other cycle) during Part II.
  Other Names: RO5509554
Drug: RO7009789 — RO7009789 will be administered IV every 3 weeks (every cycle).

SUMMARY:
This is an open-label, multicenter study designed to assess the safety, pharmacokinetics, pharmacodynamics, and therapeutic activity of emactuzumab and RO7009789 administered in combination in participants with locally advanced or metastatic solid tumors that are not amenable to standard treatment. This study will be conducted in two parts: a dose-finding stage (Part I) and an expansion stage (Part II).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status 0 or 1
* Histologically confirmed diagnosis of locally advanced, recurrent, and/or metastatic triple-negative breast cancer, ovarian cancer, gastric cancer, colorectal cancer, pancreatic cancer, melanoma, or mesothelioma
* Radiologically measurable and clinically evaluable disease as per RECIST v1.1
* Life expectancy of greater than or equal to (>/=) 16 weeks
* Ability to comply with the collection of tumor biopsies; tumors accessible for biopsy
* Adequate bone marrow, liver, cardiac, and renal function

Exclusion Criteria:

* Allergy or hypersensitivity to components of either study drug formulation
* Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening or prior radiographic assessments. Participants with radiographically stable, asymptomatic, previously irradiated lesions are eligible provided participant is >/=4 weeks beyond completion of cranial irradiation and >/=3 weeks off of corticosteroid therapy
* Participants with leptomeningeal disease; metastases to the brain stem, midbrain, pons, medulla, or within 10 millimeters (mm) of the optic apparatus (optic nerves and chiasm)
* History of human immunodeficiency virus (HIV)
* Participants with active hepatitis B, active hepatitis C, or active tuberculosis
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Up to 6 weeks from Day (D) 1 of Cycle (C) 1 (cycle = 3 weeks)

SECONDARY OUTCOMES:
Percentage of Participants with Anti-Drug Antibodies (ADAs) to Emactuzumab | Predose (PrD) (0 hours [H]) on D1 each cycle (cycle = 3 weeks) until progressive disease (PD) (up to 2 years); at 28, 44, 120 days after last dose (up to 2 years overall)
Percentage of Participants with ADAs to RO7009789 | PrD (0 H) on D1 each cycle (cycle = 3 weeks) until PD (up to 2 years); at 120 days after last dose (up to 2 years overall)
Serum Maximum Concentration (Cmax) of Emactuzumab | PrD (0 H) D1 of C1 up to 120 days after last dose (up to 2 years overall); see Outcome Measure Description for details
  PrD (0 H), end of infusion (EOI) (infusion = 90 minutes [min]), postdose [5 H] D1 of C1/C4 (cycle = 3 weeks); on D2, 5, 8, 12, 15, 19 of C1/C4; on D5, 8, 12, 17 of C2; on D2, 8, 15 of C3; PrD (0 H), EOI on D1 of C2, 3, 5 onwards until/at PD (up to 2 years); at 28, 44, 120 days after last dose (up to 2 years overall)
Serum Trough Concentration (Ctrough) of Emactuzumab | PrD (0 H) on D1 of C2 onwards (cycle = 3 weeks) until PD (up to 2 years)
Area Under the Concentration-Time Curve (AUC) of Emactuzumab | PrD (0 H) D1 of C1 up to 120 days after last dose (up to 2 years overall); see Outcome Measure Description for details
  PrD (0 H), EOI (infusion = 90 min), postdose [5 H] D1 of C1/C4; on D2, 5, 8, 12, 15, 19 of C1/C4 (cycle = 3 weeks); on D5, 8, 12, 17 of C2; on D2, 8, 15 of C3; PrD (0 H), EOI on D1 of C2, 3, 5 onwards until/at PD (up to 2 years); at 28, 44, 120 days after last dose (up to 2 years overall)
Total Clearance (CL) of Emactuzumab | PrD (0 H) D1 of C1 up to 120 days after last dose (up to 2 years overall); see Outcome Measure Description for details
  PrD (0 H), EOI (infusion = 90 min), postdose [5 H] D1 of C1/C4; on D2, 5, 8, 12, 15, 19 of C1/C4 (cycle = 3 weeks); on D5, 8, 12, 17 of C2; on D2, 8, 15 of C3; PrD (0 H), EOI on D1 of C2, 3, 5 onwards until/at PD (up to 2 years); at 28, 44, 120 days after last dose (up to 2 years overall)
Volume of Distribution at Steady State (Vss) of Emactuzumab | PrD (0 H) D1 of C1 up to 120 days after last dose (up to 2 years overall); see Outcome Measure Description for details
  PrD (0 H), EOI (infusion = 90 min), postdose [5 H] D1 of C1/C4; on D2, 5, 8, 12, 15, 19 of C1/C4 (cycle = 3 weeks); on D5, 8, 12, 17 of C2; on D2, 8, 15 of C3; PrD (0 H), EOI on D1 of C2, 3, 5 onwards until/at PD (up to 2 years); at 28, 44, 120 days after last dose (up to 2 years overall)
Accumulation Ratio of Emactuzumab | PrD (0 H) D1 of C1 up to 120 days after last dose (up to 2 years overall); see Outcome Measure Description for details
  PrD (0 H), EOI (infusion = 90 min), postdose [5 H] D1 of C1/C4; on D2, 5, 8, 12, 15, 19 of C1/C4 (cycle = 3 weeks); on D5, 8, 12, 17 of C2; on D2, 8, 15 of C3; PrD (0 H), EOI on D1 of C2, 3, 5 onwards until/at PD (up to 2 years); at 28, 44, 120 days after last dose (up to 2 years overall)
Terminal Elimination Half-Life (T1/2) of Emactuzumab | PrD (0 H) D1 of C1 up to 120 days after last dose (up to 2 years overall); see Outcome Measure Description for details
  PrD (0 H), EOI (infusion = 90 min), postdose [5 H] D1 of C1/C4; on D2, 5, 8, 12, 15, 19 of C1/C4 (cycle = 3 weeks); on D5, 8, 12, 17 of C2; on D2, 8, 15 of C3; PrD (0 H), EOI on D1 of C2, 3, 5 onwards until/at PD (up to 2 years); at 28, 44, 120 days after last dose (up to 2 years overall)
Concentration at Time of Tumor Progression (Cprog) of Emactuzumab According to Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 | At time of PD (up to 2 years)
Concentration of Emactuzumab at Time of Tumor Response (Complete or Partial Response) According to RECIST v1.1 | At time of tumor response (up to 2 years)
Concentration of Emactuzumab at Time of Infusion-Related Reaction (IRR) or Hypersensitivity Reaction | At time of IRR or hypersensitivity reaction (up to 2 years)
Cmax of RO7009789 | PrD (0 H), 15 min during infusion, EOI (infusion = 30 min), postdose (2, 4, 6 H) on D1 of C1 (cycle = 3 weeks); on D2, 3, 8 of C1; PrD (0 H), EOI on D1 of C2 onwards until/at PD (up to 2 years); at 120 days after last dose (up to 2 years overall)
Ctrough of RO7009789 | PrD (0 H) on D1 of C2 onwards (cycle = 3 weeks) until PD (up to 2 years)
AUC of RO7009789 | PrD (0 H), 15 min during infusion, EOI (infusion = 30 min), postdose (2, 4, 6 H) on D1 of C1 (cycle = 3 weeks); on D2, 3, 8 of C1; PrD (0 H), EOI on D1 of C2 onwards until/at PD (up to 2 years); at 120 days after last dose (up to 2 years overall)
CL of RO7009789 | PrD (0 H), 15 min during infusion, EOI (infusion = 30 min), postdose (2, 4, 6 H) on D1 of C1 (cycle = 3 weeks); on D2, 3, 8 of C1; PrD (0 H), EOI on D1 of C2 onwards until/at PD (up to 2 years); at 120 days after last dose (up to 2 years overall)
Vss of RO7009789 | PrD (0 H), 15 min during infusion, EOI (infusion = 30 min), postdose (2, 4, 6 H) on D1 of C1 (cycle = 3 weeks); on D2, 3, 8 of C1; PrD (0 H), EOI on D1 of C2 onwards until/at PD (up to 2 years); at 120 days after last dose (up to 2 years overall)
Accumulation Ratio of RO7009789 | PrD (0 H), 15 min during infusion, EOI (infusion = 30 min), postdose (2, 4, 6 H) on D1 of C1 (cycle = 3 weeks); on D2, 3, 8 of C1; PrD (0 H), EOI on D1 of C2 onwards until/at PD (up to 2 years); at 120 days after last dose (up to 2 years overall)
T1/2 of RO7009789 | PrD (0 H), 15 min during infusion, EOI (infusion = 30 min), postdose (2, 4, 6 H) on D1 of C1 (cycle = 3 weeks); on D2, 3, 8 of C1; PrD (0 H), EOI on D1 of C2 onwards until/at PD (up to 2 years); at 120 days after last dose (up to 2 years overall)
Total Tumor-Associated Macrophages (TAMs) in Paired-Tumor Biopsies | Baseline; on D1 of C2 (cycle = 3 weeks); and optionally at time of PD (up to 2 years)
Total Dermal Macrophages in Paired-Skin Biopsies | Baseline; on D1 of C2 (cycle = 3 weeks); and optionally at time of PD (up to 2 years)
Levels of Functional Tumor-Infiltrating Lymphocytes | Baseline; on D1 of C2 (cycle = 3 weeks); and optionally at time of PD (up to 2 years)
Circulating Colony-Stimulating Factor (CSF)-1 Serum Levels | Baseline; on D2, 5, 8, 15 of C1 (cycle = 3 weeks); on D2, 5, 15 of C3; PrD (+/- 1 day) on D1 of each cycle until/at PD (up to 2 years); at 44, 120 days after last dose (up to 2 years overall)
Total Monocyte Count in Peripheral Blood | Baseline; on D2, 5, 8, 15 of C1/C3 (cycle = 3 weeks); PrD (+/- 1 day) on D1 of each cycle until/at PD (up to 2 years); at 44, 120 days after last dose (up to 2 years overall)
Total Dendritic Cell Count in Peripheral Blood | Baseline; on D2, 5, 8, 15 of C1/C3 (cycle = 3 weeks); PrD (+/- 1 day) on D1 of each cycle until/at PD (up to 2 years); at 44, 120 days after last dose (up to 2 years overall)
Circulating Cluster of Differentiation (CD) 4 T Cell Count in Peripheral Blood | Baseline; on D2, 5, 8, 15 of C1/C3 (cycle = 3 weeks); PrD (+/- 1 day) on D1 of each cycle until/at PD (up to 2 years); at 44, 120 days after last dose (up to 2 years overall)
Circulating CD8 T Cell Count in Peripheral Blood | Baseline; on D2, 5, 8, 15 of C1/C3 (cycle = 3 weeks); PrD (+/- 1 day) on D1 of each cycle until/at PD (up to 2 years); at 44, 120 days after last dose (up to 2 years overall)
Circulating B Cell Count in Peripheral Blood | Baseline; on D2, 5, 8, 15 of C1/C3 (cycle = 3 weeks); PrD (+/- 1 day) on D1 of each cycle until/at PD (up to 2 years); at 44, 120 days after last dose (up to 2 years overall)
Metabolic Response of Target Lesions Assessed as the Change in Maximum Standardized Uptake Value (SUVmax) on [18F]-Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) | Baseline; on D15 of C1; PrD (+/- 4 days) on D1 of C3 (cycle = 3 weeks)
Percentage of Participants by Best Overall Response as Assessed by RECIST v1.1 | Baseline; every 6 weeks until PD (up to 2 years); at 28 days after last dose (up to 2 years overall)
Percentage of Participants with Overall Response as Assessed by RECIST v1.1 | Baseline; every 6 weeks until PD (up to 2 years); at 28 days after last dose (up to 2 years overall)
Progressive-Free Survival (PFS) as Assessed by RECIST v1.1 | From Baseline until death or PD; assessed every 6 weeks (up to 2 years overall)
Duration of Response (DOR) as Assessed by RECIST v1.1 | From OR until PD; assessed every 6 weeks (up to 2 years overall)
Percentage of Participants with Clinical Benefit as Assessed by RECIST v1.1 | Baseline; every 6 weeks until PD (up to 2 years); at 28 days after last dose (up to 2 years overall)
Percentage of Participants by Best Overall Response as Assessed by Modified RECIST | Baseline; every 6 weeks until PD (up to 2 years); at 28 days after last dose (up to 2 years overall)
Percentage of Participants with Overall Response as Assessed by Modified RECIST | Baseline; every 6 weeks until PD (up to 2 years); at 28 days after last dose (up to 2 years overall)
Progressive-Free Survival (PFS) as Assessed by Modified RECIST | From Baseline until death or PD; assessed every 6 weeks (up to 2 years overall)
Duration of Response (DOR) as Assessed by Modified RECIST | From OR until PD; assessed every 6 weeks (up to 2 years overall)
Percentage of Participants with Clinical Benefit as Assessed by Modified RECIST | Baseline; every 6 weeks until PD (up to 2 years); at 28 days after last dose (up to 2 years overall)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University Pennsylvania Hospital, Philadelphia, Pennsylvania
- Cliniques Universitaires St-Luc, Brussels, Belgium
- France (3):
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy; Sitep, Villejuif

REFERENCES:
- [Derived] Machiels JP, Gomez-Roca C, Michot JM, Zamarin D, Mitchell T, Catala G, Eberst L, Jacob W, Jegg AM, Cannarile MA, Watson C, Babitzki G, Korski K, Klaman I, Teixeira P, Hoves S, Ries C, Meneses-Lorente G, Michielin F, Christen R, Ruttinger D, Weisser M, Delord JP, Cassier P. Phase Ib study of anti-CSF-1R antibody emactuzumab in combination with CD40 agonist selicrelumab in advanced solid tumor patients. J Immunother Cancer. 2020 Oct;8(2):e001153. doi: 10.1136/jitc-2020-001153. PMID 33097612